CLINICAL TRIAL: NCT02926976
Title: The Optimal Treatment for Treatment-resistant Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The optimal treatment for TRS
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Clozapine; Aripiprazole; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- risperidone with clozapine (Active Comparator): risperidone, dosage form: 1 mg, dosage and frequency:3.0~6.0 mg/d; clozapine, dosage and frequency:300~600 mg/d; duration: 8 weeks
  Interventions: Drug: Risperidone with Clozapine
- aripiprazole with clozapine (Active Comparator): aripiprazole, dosage form: 5 mg, dosage and frequency:15~30 mg/day; clozapine, dosage and frequency:300~600 mg/d; duration: 8 weeks
  Interventions: Drug: Aripiprazole with Clozapine
- sodium valproate with clozapine (Active Comparator): sodium valproate, dosage form: 250 mg, dosage and frequency:600~1200 mg/day; clozapine, dosage and frequency:300~600 mg/d; duration: 3 months.
  Interventions: Drug: sodium valproate with Clozapine
- clozapine (Active Comparator): only clozapine, dosage and frequency:300~600 mg/d;
  Interventions: Device: clozapine
- Modified electroconvulsive therapy with clozapine (Active Comparator): 10 times MECT for 4 weeks, if the PANSS reductive ratio is less 20% in the end of 8th week by the using of risperidone with clozapine, aripiprazole with clozapine, sodium valproate with clozapine, or clozapine.
  Interventions: Device: modified electroconvulsive therapy(MECT) with Clozapine
- Magnetic seizure therapy with clozapine (Active Comparator): 10 times MST for 4 weeks, if the PANSS reductive ratio is less 20% in the end of 8th week by the using of risperidone with clozapine, aripiprazole with clozapine, sodium valproate with clozapine, or clozapine.
  Interventions: Device: Magnetic seizure therapy(MST) with Clozapine

INTERVENTIONS:
Drug: Risperidone with Clozapine — Risperidone may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia
  Other Names: Risperidone Tablet
  Arms: risperidone with clozapine
Drug: Aripiprazole with Clozapine — Aripiprazole may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia
  Other Names: Aripiprazole Tablets
  Arms: aripiprazole with clozapine
Drug: sodium valproate with Clozapine — sodium valproate may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia
  Other Names: Valproate
  Arms: sodium valproate with clozapine
Device: modified electroconvulsive therapy(MECT) with Clozapine — modified electroconvulsive therapy(MECT) may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia
  Arms: Modified electroconvulsive therapy with clozapine
Device: Magnetic seizure therapy(MST) with Clozapine — Magnetic seizure therapy(MST) may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia
  Arms: Magnetic seizure therapy with clozapine
Device: clozapine — clozapine may be used in the treatment of treatment-resistant schizophrenia
  Arms: clozapine

SUMMARY:
The Optimal Treatment for Treatment-resistant Schizophrenia

DETAILED DESCRIPTION:
To explore the curative effect and safety of Risperidone，aripiprazole，sodium valproate，modified electroconvulsive therapy(MECT), or Magnetic seizure therapy(MST) with Clozapine in the treatment of treatment-resistant schizophrenia， and to provide the basis for clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of schizophrenia according to DSM-V
* 18～60 years old
* 2 prior failed treatment trials with 2 different antipsychotics at doses of at least 600 mg/day chlorpromazine equivalents, each of at least 6 weeks duration;
* Signed an informed consent

Exclusion Criteria:

* patients to be diagnosed according to DSM-V for substance abused, development delayed
* suffering from serious physical disease and can not accept the treatment
* MST contraindications: intracranial metal substance, with heart pacemakers and cochlear implants, intracranial pressure
* allergic to risperidone ,aripiprazole, or sodium valproate
* Participated in any clinical subject within 30 days
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale [PANSS] | At baseline, 4th week, 8th week,12th week

SECONDARY OUTCOMES:
Change from baseline in clinical global impression [CGI] | At baseline, 4th week, 8th week,12th week
Change from baseline in Simpson-Angus Scale [SAS] | At baseline, 4th week, 8th week,12th week
Change from baseline in Abnormal Involuntary Movement Scale[AIMS] | At baseline, 4th week, 8th week,12th week

CONTACTS AND LOCATIONS:
Locations (1):
- DTliu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No